CLINICAL TRIAL: NCT02990962
Title: The Long-term Effect of Perineural Injection Therapy Versus Steroid in Patients With Carpal Tunnel Syndrome
Brief Title: The Effect of Perineural Injection Therapy Versus Steroid in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending physician of physical medicine and rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIT for CTS
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: perineural injection; ultrasound-guided; dextrose; steroid
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perineural injection with 5% dextrose (Experimental): Ultrasound-guided perineural injection with 5% Dextrose (5cc) between carpal tunnel and median nerve.
  Interventions: Drug: 5% dextrose
- Perineural injection with steroid (Active Comparator): Ultrasound-guided perineural injection with 1cc 2% Xylocaine+4cc Triamcinolone (40mg) between carpal tunnel and median nerve.
  Interventions: Drug: 1cc 2% Xylocaine+4cc Triamcinolone (40mg)

INTERVENTIONS:
Drug: 5% dextrose — Ultrasound-guided perineural injection with 5% dextrose (5cc) between carpal tunnel and surrounding median nerve with hydrodissection.
  Arms: Perineural injection with 5% dextrose
Drug: 1cc 2% Xylocaine+4cc Triamcinolone (40mg) — Ultrasound-guided perineural injection with1cc 2% Xylocaine+4cc Triamcinolone (40mg) between carpal tunnel and surrounding median nerve with hydrodissection.
  Arms: Perineural injection with steroid

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. Rather than other progressive disease, CTS is characterized by remission and recurrence. Although many conservative managements of CTS, the effectiveness of these methods is insignificant or only persist for a short duration including steroid injection. Recently, the ultrasound-guided perineural injection with 5% dextrose was widely used for entrapment neuropathy with positive benefit. The investigators design a randomized, double-blind, controlled trail to assess the effect of ultrasound-guided perineural injection with 5% dextrose in patients with CTS and compared with steroid injection.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients of clinically diagnosed with CTS were randomized into intervention and control group. Participants in intervention group received one-session ultrasound-guided perineural injection with 5% dextrose and control group received one-session ultrasound-guided perineural injection with steroid. No additional treatment after injection through the study period. The primary outcome is visual analog scale (VAS) and secondary outcomes include Boston Carpal Tunnel Syndrome Questionnaire (BCTQ), cross-sectional area (CSA) of the median nerve, sensory nerve conduction velocity of the median nerve, and finger pinch strength. The evaluation was performed pretreatment as well as on the 2nd week, 1st, 2nd, 3rd and 6 month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-85 year-old.
* Diagnosis was confirmed using an electrophysiological study and ultrasonography

Exclusion Criteria:

Cancer

* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st, 2nd, 3rd and 6 month after the treatment. | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 2nd week, 1st, 2nd, 3rd and 6 month after the treatment. | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  Using the Boston Carpal Tunnel Syndrome Questionnaire to measure the symptoms and functional status before treatment and multiple time frame after treatment
Change from baseline of cross-sectional area of the median nerve on 2nd week, 1st, 2nd, 3rd and 6 month after the treatment. | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve.
Change from baseline of nerve conduction velicity on 2nd week, 1st, 2nd, 3rd and 6 month after the treatment. | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  Nerve motor conduction velocity of the ulnar nerve before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Mulvaney SW. Ultrasound-guided percutaneous neuroplasty of the lateral femoral cutaneous nerve for the treatment of meralgia paresthetica: a case report and description of a new ultrasound-guided technique. Curr Sports Med Rep. 2011 Mar-Apr;10(2):99-104. doi: 10.1249/JSR.0b013e3182110096. PMID 21623291
- [Result] Tsui BC, Wagner A, Finucane B. Electrophysiologic effect of injectates on peripheral nerve stimulation. Reg Anesth Pain Med. 2004 May-Jun;29(3):189-93. doi: 10.1016/j.rapm.2004.02.002. PMID 15138901
- [Result] Tsui BCH, Kropelin B. The electrophysiological effect of dextrose 5% in water on single-shot peripheral nerve stimulation. Anesth Analg. 2005 Jun;100(6):1837-1839. doi: 10.1213/01.ANE.0000153020.84780.A5. PMID 15920223
- [Result] Girlanda P, Dattola R, Venuto C, Mangiapane R, Nicolosi C, Messina C. Local steroid treatment in idiopathic carpal tunnel syndrome: short- and long-term efficacy. J Neurol. 1993;240(3):187-90. doi: 10.1007/BF00857526. PMID 8482993
- [Result] Armstrong T, Devor W, Borschel L, Contreras R. Intracarpal steroid injection is safe and effective for short-term management of carpal tunnel syndrome. Muscle Nerve. 2004 Jan;29(1):82-8. doi: 10.1002/mus.10512. PMID 14694502